CLINICAL TRIAL: NCT03191721
Title: Effects of a Toothpaste Containing 0.3% Triclosan in the Maintenance Phase of Peri-implantitis Treatment.
Brief Title: Triclosan Toothpaste in the Maintenance Phase of Peri-implantitis Treatment.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Guarulhos (Other)
Collaborators: Universidade Estadual de Maringá (Other)
Responsible Party: Principal Investigator, Belén Retamal-Valdes, DDS, MSc, PhD Student, University of Guarulhos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE - 0007.0.132.000-10
Record Dates: First submitted 2017-06-08; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Peri-Implantitis; Periodontal Diseases
Keywords: Peri-implantitis; Triclosan; Toothpastes; Therapeutics; Periodontal Diseases; Periodontitis; Dentifrices
MeSH Terms: conditions — Peri-Implantitis; Periodontal Diseases; Periodontitis | interventions — Periodontal Index; Triclosan; Fluorides; Maintenance

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test: Triclosan toothpaste (Experimental): To brush twice a day with a toothpaste containing 0.3% triclosan and 1450 ppm sodium fluoride in a regular maintenance program for 24 months.
  Two months earlier, subjects received Surgical anti-infective therapy for implants with peri-implantitis, periodontal treatment and oral hygiene instruction.
  Interventions: Procedure: Surgical anti-infective therapy; Procedure: Periodontal treatment; Procedure: Oral Hygiene Instruction; Drug: Triclosan toothpaste; Procedure: Regular maintenance program
- Control: Fluoride toothpaste (Placebo Comparator): To brush twice a day with a toothpaste containing 1450 ppm sodium monofluorphosphate in a regular maintenance program for 24 months.
  Two months earlier, subjects received Surgical anti-infective therapy for implants with peri-implantitis, periodontal treatment and oral hygiene instruction.
  Interventions: Procedure: Surgical anti-infective therapy; Procedure: Periodontal treatment; Procedure: Oral Hygiene Instruction; Drug: Fluoride toothpaste; Procedure: Regular maintenance program

INTERVENTIONS:
Procedure: Surgical anti-infective therapy — Two months before randomization, implants with peri-implantitis received surgical anti-infective therapy. After local anesthesia (2% lidocaine with 1:100,000 epinephrine), intrasulcular incisions were done and buccal and lingual full-thickness flaps were dissected. Granulation tissue was removed to expose the implant threads and bone defect. To remove biofilm and calculus, the implant surface was scaled with teflon curettes and decontaminated with bicarbonate jet (Jet Sonic System). The flap was repositioned in the original position and stabilized with interrupted sutures, which were removed after 10 days
  Other Names: Pre-baseline phase - surgery
Procedure: Periodontal treatment — Two months before randomization, all subjects received full-mouth supragingival plaque removal and scaling and root planing (SRP), as needed. The SRP was performed in four to six appointments lasting approximately 1 h each, using manual curettes (Hu-Friedy, Chicago, IL, USA) and ultrasonic device (Cavitron Select SPC, Dentsply professional, York, PA, USA) under local anesthesia. The deep sites were scaled throughout the first week and treatment of the entire oral cavity was completed in 14 days.
  Other Names: Pre-baseline phase - SRP
Procedure: Oral Hygiene Instruction — Delivery of a soft bristle adult toothbrush (Colgate Palmolive, Brazil), dental floss (Colgate Palmolive, Brazil), and interdental toothbrushes (Colgate Palmolive, Brazil) , according to their individual needs at pre-baseline, baseline, 3, 6, 12, 18 and 24 months. Information was given about the importance of keeping an excellent oral hygiene over the course of the study. The subjects were instructed to brush their teeth for one minute twice a day (morning and evening) using only the toothbrush and toothpaste provided.
  Other Names: OHI
Drug: Triclosan toothpaste — Dental brushing with a toothpaste containing 0.3% triclosan and 1450 ppm sodium fluoride in a regular maintenance program for 24 months.
  Other Names: Triclosan
  Arms: Test: Triclosan toothpaste
Drug: Fluoride toothpaste — Dental brushing with a toothpaste containing 1450 ppm sodium monofluorphosphate in a regular maintenance program for 24 months.
  Other Names: Fluoride
  Arms: Control: Fluoride toothpaste
Procedure: Regular maintenance program — OHI, supragingival and subgingival biofilm removal from teeth and implants, and oral prophylaxis. If the examiner suspected of peri-implant disease progression, periapical radiographs were taken. If the implant showed ≥ 2 mm of bone loss, it was withdrawn from the study to receive additional treatment (e.g. another surgery procedure). Implants showing severe disease progression associated with mobility were removed. Maintenance visits were performed every 3 months.
  Other Names: Maintenance

SUMMARY:
The aim of this study was to evaluate the effects of a dentifrice containing 0.3% triclosan on periodontal and peri-implant parameters in patients, with or without periodontitis, treated for peri-implantitis and that were enrolled in a maintenance phase for two years.

DETAILED DESCRIPTION:
Although dental implants have a high success rate, the prevalence of peri-implantitis has been rising worldwide. Similarly to periodontitis, peri-implantis are complex infections caused by oral pathogens that colonize the oral cavity tissues. Then, several anti-infective treatments have been proposed to treat peri-implantitis. Although an ideal and definitive therapy has not yet been established, one of the most commonly used protocols is the open-flap mechanical decontamination of the implant surfaces. Nonetheless, it has been well established that after the active treatment phase, it is essential that patients enter a maintenance phase, similarly to that followed by patients who have had periodontitis. One of the main risk indicators for peri-implantitis is poor oral hygiene, so the maintenance phase should include strict control of the supra and submucosal biofilms. Several methods, including the use of dental and interdental brushes, are usually recommended for the mechanical control of biofilm accumulated in implant surfaces; however, many patients are not able to effectively remove this biofilm. Thus, the use of a chemical adjunct to traditional mechanical methods during the maintenance phase of peri-implantitis treatment could improve the long term stability of dental implants. Among the several antimicrobial agents used to control biofilm accumulation in the oral cavity, triclosan is one of the most effective. Therefore, the aim of this study was to evaluate the effects of a dentifrice containing 0.3% triclosan on periodontal and peri-implant parameters in patients, with or without periodontitis, treated for peri-implantitis and that were enrolled in a maintenance phase for two years. Subjects presenting at least one implant with peri-implantitis, received surgical anti-infective therapy consisting of mechanical debridement of the implant surfaces with scalers and sodium bicarbonate jet were entered into the study. Sixty days later (baseline), subjects were randomized into two groups: (i) brushing with a toothpaste containing 0.3% triclosan + 1450 ppm fluoride (test) or (ii) brushing with a toothpaste containing 1450 ppm fluoride (control). Subjects received clinical and microbiological monitoring at baseline, 3, 6, 12, 18 and 24 months post-therapy. 102 subjects were enrolled (test, n= 48; control, n=54) in the study. The results for peri-implant parameters showed that the control group had loss of relative clinical attachment level (CAL) over the course of the study (p<0.05) while the test group showed stability for this parameter. The difference between groups for CAL change between baseline and 24 months (0.55 mm) was statistically significant (primary outcome variable). The red complex pathogens were only reduced in the test group at 24 months. The periodontal parameters results showed that the test group (n=39) had a greater reduction in the percentage of sites exhibiting bleeding on probing and lower levels of plaque in comparison with the control group (n=49) after 24 months of brushing with the assigned toothpastes (p<0.05). The mean percentage of sites with probing depth ≥ 5mm was reduced over the course of the study only in the test group (p<0.05). The data of the present study showed that a toothpaste containing 0.3% triclosan was more effective than a regular fluoride toothpaste in maintaining peri-implant clinical stability and a more beneficial subgingival microbial profile in subjects with or without a history of periodontitis, that have been treated for peri-implantitis and were enrolled in a regular maintenance program for 2 years. In addition, a toothpaste containing 0.3% triclosan was more effective in maintaining a healthier periodontal environment around natural teeth.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-70 years;
* general good health;
* minimum of 1 dental implant in function for at least one year with untreated peri-implantitis defined as: probing depth (PD) ≥ 5 mm, bleeding on probing (BOP) or suppuration, radiographic bone loss involving 2 mm from the upper border of the intrabony portion of the implant.

Exclusion Criteria:

* untreated periodontitis (defined as ≥ 6 sites with PD ≥ 5 mm);
* periodontal treatment within three months prior to entering the study;
* inability to perform proper supragingival plaque control (e.g. due to improper prosthesis design or lack of skills);
* diabetes;
* pregnancy;
* nursing;
* history of allergies to triclosan, fluoride or any other ingredient of oral care products;
* alcohol or drug abuse;
* any systemic diseases that could affect post-operative healing;
* any systemic diseases that required antibiotic premedication for routine dental therapy;
* long-term use of mouthrinses, anti-inflammatory medications or any other drug that could interfere with the study outcomes within three months prior to entering the study;
* antibiotics use within six months prior to entering the study;
* participation in any other clinical study within three months prior to entering the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level (CAL) at 24 months. | 24 months
  Difference between groups for the change in Clinical Attachment Level (CAL) from baseline to 24 months.

SECONDARY OUTCOMES:
Probing Depth (PD) ≥ 5 mm. | Baseline, 3, 6, 12, 18, 24 months.
  Number of sites with Probing Depth (PD) ≥ 5 mm, evaluated in all volunteers.
PD ≥ 6 mm. | Baseline, 3, 6, 12, 18, 24 months.
  Number of sites with PD ≥ 6 mm, evaluated in all volunteers.
PD ≥ 7 mm. | Baseline, 3, 6, 12, 18, 24 months.
  Number of sites with PD ≥ 7 mm, evaluated in all volunteers.
Full-mouth PD. | Baseline, 3, 6, 12, 18, 24 months.
  Mean of the PD evaluated in all the periodontal sites from all volunteers.
Full-mouth CAL. | Baseline, 3, 6, 12, 18, 24 months.
  Mean of the CAL evaluated in all the periodontal sites from all volunteers.
Bleeding on Probing (BOP). | Baseline, 3, 6, 12, 18, 24 months.
  Percentage of sites with bleeding on probing (BOP), evaluated in all volunteers.
Plaque accumulation. | Baseline, 3, 6, 12, 18, 24 months.
  Percentage of sites with plaque accumulation, evaluated in all volunteers.
Marginal bleeding. | Baseline, 3, 6, 12, 18, 24 months.
  Percentage of sites with marginal bleeding.
Sites gaining CAL ≥ 2mm. | Baseline - 24 months.
  Percentage of sites gaining ≥ 2mm of CAL.
Sites loosing CAL ≥ 2mm | Baseline - 24 months.
  Percentage of sites loosing ≥ 2mm of CAL
Radiographic Bone Height | Baseline, 3, 6, 12, 18, 24 months.
  Mean values of radiographic bone height
BOP reduction | Baseline - 24 months.
  Reduction in the percentage of sites exhibiting BOP.
Adverse effects | 3, 6, 12, 18, 24 months.
  Occurrence of nausea and irritability obtained through a questionnaire of adverse effects
Proportions of periodontal pathogenic bacterial species. | Baseline, 3, 6, 12, 18, 24 months.
  Proportions of periodontal pathogenic bacterial species in subgingival biofilm samples.
Counts of periodontal pathogenic bacterial species. | Baseline, 3, 6, 12, 18, 24 months.
  Proportions of periodontal pathogenic bacterial species in subgingival biofilm samples.

CONTACTS AND LOCATIONS:
Overall Officials: Magda Feres, Professor, Study Director — Guarulhos University; Bernal Stewart, Study Chair — Colgate-Palmolive Company
Locations (2):
- Brazil (2):
  - State University of Maringa, Maringa, Santa Catarina
  - Guarulhos University, Guarulhos, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
March 2017

REFERENCES:
- [Background] Cumming BR, Loe H. Consistency of plaque distribution in individuals without special home care instruction. J Periodontal Res. 1973;8(2):94-100. doi: 10.1111/j.1600-0765.1973.tb00756.x. No abstract available. PMID 4267951
- [Background] de Mendonca AC, Santos VR, Cesar-Neto JB, Duarte PM. Tumor necrosis factor-alpha levels after surgical anti-infective mechanical therapy for peri-implantitis: a 12-month follow-up. J Periodontol. 2009 Apr;80(4):693-9. doi: 10.1902/jop.2009.080521. PMID 19335091
- [Background] Derks J, Schaller D, Hakansson J, Wennstrom JL, Tomasi C, Berglundh T. Effectiveness of Implant Therapy Analyzed in a Swedish Population: Prevalence of Peri-implantitis. J Dent Res. 2016 Jan;95(1):43-9. doi: 10.1177/0022034515608832. PMID 26701919
- [Background] Derks J, Tomasi C. Peri-implant health and disease. A systematic review of current epidemiology. J Clin Periodontol. 2015 Apr;42 Suppl 16:S158-71. doi: 10.1111/jcpe.12334. PMID 25495683
- [Background] Duarte PM, de Mendonca AC, Maximo MB, Santos VR, Bastos MF, Nociti FH. Effect of anti-infective mechanical therapy on clinical parameters and cytokine levels in human peri-implant diseases. J Periodontol. 2009 Feb;80(2):234-43. doi: 10.1902/jop.2009.070672. PMID 19186963
- [Background] Figuero E, Graziani F, Sanz I, Herrera D, Sanz M. Management of peri-implant mucositis and peri-implantitis. Periodontol 2000. 2014 Oct;66(1):255-73. doi: 10.1111/prd.12049. PMID 25123773
- [Background] Heitz-Mayfield LJ, Lang NP. Comparative biology of chronic and aggressive periodontitis vs. peri-implantitis. Periodontol 2000. 2010 Jun;53:167-81. doi: 10.1111/j.1600-0757.2010.00348.x. PMID 20403112
- [Background] Heitz-Mayfield LJ, Mombelli A. The therapy of peri-implantitis: a systematic review. Int J Oral Maxillofac Implants. 2014;29 Suppl:325-45. doi: 10.11607/jomi.2014suppl.g5.3. PMID 24660207
- [Background] Heitz-Mayfield LJA, Salvi GE, Mombelli A, Faddy M, Lang NP. Anti-infective surgical therapy of peri-implantitis. A 12-month prospective clinical study. Clin Oral Implants Res. 2012 Feb;23(2):205-210. doi: 10.1111/j.1600-0501.2011.02276.x. Epub 2011 Aug 9. PMID 22092831
- [Background] Heitz-Mayfield LJA, Salvi GE, Mombelli A, Loup PJ, Heitz F, Kruger E, Lang NP. Supportive peri-implant therapy following anti-infective surgical peri-implantitis treatment: 5-year survival and success. Clin Oral Implants Res. 2018 Jan;29(1):1-6. doi: 10.1111/clr.12910. Epub 2016 Jun 23. PMID 27335316
- [Background] Lindhe J, Meyle J; Group D of European Workshop on Periodontology. Peri-implant diseases: Consensus Report of the Sixth European Workshop on Periodontology. J Clin Periodontol. 2008 Sep;35(8 Suppl):282-5. doi: 10.1111/j.1600-051X.2008.01283.x. PMID 18724855
- [Background] Mombelli A, Muller N, Cionca N. The epidemiology of peri-implantitis. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:67-76. doi: 10.1111/j.1600-0501.2012.02541.x. PMID 23062130
- [Background] Panagakos FS, Volpe AR, Petrone ME, DeVizio W, Davies RM, Proskin HM. Advanced oral antibacterial/anti-inflammatory technology: A comprehensive review of the clinical benefits of a triclosan/copolymer/fluoride dentifrice. J Clin Dent. 2005;16 Suppl:S1-19. PMID 16583598
- [Background] Socransky SS, Smith C, Martin L, Paster BJ, Dewhirst FE, Levin AE. "Checkerboard" DNA-DNA hybridization. Biotechniques. 1994 Oct;17(4):788-92. PMID 7833043
- [Background] Mestnik MJ, Feres M, Figueiredo LC, Duarte PM, Lira EA, Faveri M. Short-term benefits of the adjunctive use of metronidazole plus amoxicillin in the microbial profile and in the clinical parameters of subjects with generalized aggressive periodontitis. J Clin Periodontol. 2010 Apr;37(4):353-65. doi: 10.1111/j.1600-051X.2010.01538.x. PMID 20447259
- [Background] Tonetti MS, Eickholz P, Loos BG, Papapanou P, van der Velden U, Armitage G, Bouchard P, Deinzer R, Dietrich T, Hughes F, Kocher T, Lang NP, Lopez R, Needleman I, Newton T, Nibali L, Pretzl B, Ramseier C, Sanz-Sanchez I, Schlagenhauf U, Suvan JE. Principles in prevention of periodontal diseases: Consensus report of group 1 of the 11th European Workshop on Periodontology on effective prevention of periodontal and peri-implant diseases. J Clin Periodontol. 2015 Apr;42 Suppl 16:S5-11. doi: 10.1111/jcpe.12368. PMID 25639948
- [Background] Xu T, Deshmukh M, Barnes VM, Trivedi HM, Du-Thumm L, Richter R, Cummins D. Analysis of the antibacterial activity and plaque control benefit of colgate total dentifrice via clinical evaluation and real-time polymerase chain reaction. J Clin Dent. 2005;16(4):117-22. PMID 16583596
- [Background] Zitzmann NU, Berglundh T. Definition and prevalence of peri-implant diseases. J Clin Periodontol. 2008 Sep;35(8 Suppl):286-91. doi: 10.1111/j.1600-051X.2008.01274.x. PMID 18724856
- [Result] Fine DH, Furgang D, Bonta Y, DeVizio W, Volpe AR, Reynolds H, Zambon JJ, Dunford RG. Efficacy of a triclosan/NaF dentifrice in the control of plaque and gingivitis and concurrent oral microflora monitoring. Am J Dent. 1998 Dec;11(6):259-70. PMID 10477976
- [Result] Haraszthy VI, Zambon JJ, Sreenivasan PK. Evaluation of the antimicrobial activity of dentifrices on human oral bacteria. J Clin Dent. 2010;21(4):96-100. PMID 21269037
- [Result] Ramberg P, Lindhe J, Botticelli D, Botticelli A. The effect of a triclosan dentifrice on mucositis in subjects with dental implants: a six-month clinical study. J Clin Dent. 2009;20(3):103-7. PMID 19711612
- [Result] Riley P, Lamont T. Triclosan/copolymer containing toothpastes for oral health. Cochrane Database Syst Rev. 2013 Dec 5;2013(12):CD010514. doi: 10.1002/14651858.CD010514.pub2. PMID 24310847
- [Result] Rosling B, Wannfors B, Volpe AR, Furuichi Y, Ramberg P, Lindhe J. The use of a triclosan/copolymer dentifrice may retard the progression of periodontitis. J Clin Periodontol. 1997 Dec;24(12):873-80. doi: 10.1111/j.1600-051x.1997.tb01205.x. PMID 9442423
- [Result] Sreenivasan PK, Vered Y, Zini A, Mann J, Kolog H, Steinberg D, Zambon JJ, Haraszthy VI, da Silva MP, De Vizio W. A 6-month study of the effects of 0.3% triclosan/copolymer dentifrice on dental implants. J Clin Periodontol. 2011 Jan;38(1):33-42. doi: 10.1111/j.1600-051X.2010.01617.x. Epub 2010 Sep 13. PMID 20831669
- [Derived] Stewart B, Shibli JA, Araujo M, Figueiredo LC, Panagakos F, Matarazzo F, Mairink R, Onuma T, Faveri M, Retamal-Valdes B, Feres M. Effects of a toothpaste containing 0.3% triclosan in the maintenance phase of peri-implantitis treatment: 2-Year randomized clinical trial. Clin Oral Implants Res. 2018 Oct;29(10):973-985. doi: 10.1111/clr.13363. PMID 30328176